CLINICAL TRIAL: NCT03557762
Title: The SEAMLESS Study: A Clinical Trial Evaluation of a SmartphonE App-based MindfuLnEss Intervention for Cancer SurvivorS
Brief Title: The SEAMLESS Study: Smartphone App-based Mindfulness for Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Linda E. Carlson, Enbridge Research Chair in Psychosocial Oncology, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HREBA.CC-18-0029
Record Dates: First submitted 2018-06-04; First posted 2018-06-15 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Cancer; Psychological
Keywords: Cancer survivors; Smartphone app; Mindfulness
MeSH Terms: conditions — Neoplasms | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Mindfulness (Experimental): A 4 week smartphone app-based mindfulness intervention program with in-app activities for 20-30 minutes every day, with a minimum of 4 days of activity in a week.
  Interventions: Behavioral: Mindfulness
- Waitlist Control Mindfulness (Other): No intervention for 4 weeks, after which there will be assessments immediately post-waiting and at 3 months post-baseline. After this, participants will get the same 4 week smartphone app-based mindfulness intervention program.
  Interventions: Behavioral: Mindfulness

INTERVENTIONS:
Behavioral: Mindfulness — A psychological behavioral intervention that trains participants in mindfulness techniques, which involves achieving a moment-to-moment non-judgmental awareness of their internal psychosocial-emotional state, through meditation and gentle mindful movements.

SUMMARY:
Smartphone app-based health interventions are an innovative way to deliver psychosocial cancer-care. In the SEAMLESS study, the investigators aim to evaluate a 4 week smartphone app-based mind-body intervention (MBI) in cancer survivors post-treatment. This is a randomized controlled trial, with a waitlist control group. Participants will be assigned to either receive the intervention immediately after enrollment or will need to wait for 3 months to receive the intervention.

DETAILED DESCRIPTION:
BACKGROUND Cancer patients who are in the transition phase to survivorship after completing their final treatments need psychosocial interventions to manage stressors such as anxiety, depression, and fear of cancer recurrence. Smartphone app-based health interventions are an innovative way to deliver psychosocial cancer-care. In the SEAMLESS study, the investigators aim to evaluate an app-based mind-body intervention (MBI) in cancer survivors.

The need for psychosocial interventions for cancer survivors has been highlighted by the Institute of Medicine in their landmark survivorship report appropriately titled, "Lost in Transition." Cancer survivors are often unable to participate in face-to-face interventions because of difficulties such as compromised immunity, treatment-related side-effects, scheduling conflicts and geography. A smartphone-app based MBI can overcome several such difficulties, since patients can participate at their own convenience without the burden of travel and scheduling classes.

INTERVENTION DESIGN The AM smartphone app supports personalized mindfulness practices through lessons and personalized guided-meditation playlists; AM reportedly reduced anxiety in a study with college students. AM interprets its users' emotional state, e.g. angry, elated, from a user-inputted digital emotion-mapping board; and heart-rate data through algorithms that analyze facial bio-signals. The SEAMLESS study is a randomized wait-list controlled trial, which will evaluate AM's effectiveness for reducing stress (primary outcome), anxiety, depression, fatigue and fear of cancer recurrence in cancer survivors who have completed all treatments for 2 weeks or more. Outcomes will be assessed online using validated PROMIS measures at 1) baseline, 2) mid-point 3) immediately post-intervention, 4&5) 3 and 6 months follow-up post-baseline.

SIGNIFICANCE Cancer-care providers are uncertain about the efficacy of app-based interventions for patients, which are available in great supply in today's digital world. This study will provide rigorously evaluated efficacy data for an app-based MBI for cancer survivors, which if helpful, could be made easily available for psychosocial care at cancer centers worldwide.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women over the age of 18
2. Diagnosed with any type of cancer (stage I-III)
3. Completed active treatment (i.e. surgery, chemotherapy, radiation therapy) at least 4 months previously (ongoing hormonal therapies, AIs, tamoxifen, herceptin are not exclusionary)
4. Have access to a smartphone with data connection; in case patients' do not have a data plan or an insufficient data plan with their smart phone, we will pay for their data connection (up to 0.5GB/month)
5. Willing to devote 20-30 mins of time to do the mindfulness meditations and practices every day
6. Sufficient cognitive function to participate in the smartphone app-based intervention
7. Ability to speak and write English sufficiently to complete questionnaires

Exclusion Criteria:

1. Metastatic patients and those with ongoing chemotherapy (metastatic patients may not be stable enough to participate in the interventions and follow-up assessments).
2. Cognitive impairment that would interfere with completing questionnaires or the intervention.
3. Suffering from current Major Depressive Disorder, Bipolar Disorder or other psychiatric disorder that would interfere with the ability to participate.
4. Practicing smartphone app-based mindfulness more than or equal to once a week

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2020-01-06 (Actual); Study Completion 2020-08-06 (Actual)

PRIMARY OUTCOMES:
Symptoms of Stress | 3 months
  Calgary - Symptoms of Stress Inventory (C-SOSI)

SECONDARY OUTCOMES:
Fear of Cancer Recurrence | 3 months
  Fear of Cancer Recurrence Inventory (FCRI)
Anxiety - PROMIS | 3 months
  PROMIS- Cancer Bank v1.0 - Anxiety
Depression - PROMIS | 3 months
  PROMIS- Cancer Bank v1.0 - Depression
Fatigue - PROMIS | 3 months
  PROMIS- Cancer Bank v1.0 - Fatigue
Physical Function - PROMIS | 3 months
  PROMIS- Cancer Bank v1.1 - Physical Function
App-based User Data | 3 months
  Users' self-reported stress, biometrics and engagement

CONTACTS AND LOCATIONS:
Overall Officials: Linda Carlson, PhD, Principal Investigator — University of Calgary
Locations (1):
- Psychosocial Oncology, Cancer Control Alberta, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD